CLINICAL TRIAL: NCT05631626
Title: A Phase 3, Dose-Optimized, Randomized, Double-Blind, Placebo-Controlled, Single-Center, Parallel Efficacy and Safety Laboratory Classroom Study in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD) Using CTx-1301 (Dexmethylphenidate)
Brief Title: Phase 3 Efficacy and Safety Study in Adults With ADHD Using CTx-1301.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cingulate Therapeutics (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTx-1301-022
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-06

CONDITIONS: ADHD; ADHD - Combined Type; Attention Deficit Hyperactivity Disorder Combined; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 25mg CTx-1301 (Dexmethylphenidate tablet) (Active Comparator): All subjects will be titrated to their optimal dose during the dose-optimization phase. The starting dose for all subjects at Day 0 is 25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 25mg
- 37.5mg CTx-1301 (Dexmethylphenidate tablet) (Active Comparator): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 25mg, 37.5mg, or 50mg . Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 37.5mg
- 50mg CTx-1301 (Dexmethylphenidate tablet) (Active Comparator): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 25mg, 37.5mg, or 50mg . Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 50mg
- Placebo (Placebo Comparator): Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTx-1301 - Dexmethylphenidate 25mg — 25mg CTx-1301 (Dexmethylphenidate tablet)
  Other Names: All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 25mg, 37.5mg, or 50mg of CTx-1301.
  Arms: 25mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 37.5mg — 37.5mg CTx-1301 (Dexmethylphenidate tablet)
  Other Names: All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 25mg, 37.5mg, or 50mg of CTx-1301.
  Arms: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 50mg — 50mg CTx-1301 (Dexmethylphenidate tablet)
  Other Names: All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 25mg, 37.5mg, or 50mg of CTx-1301.
  Arms: 50mg CTx-1301 (Dexmethylphenidate tablet)
Drug: Placebo — Placebo
  Other Names: Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomized phase.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of CTx-1301 in adults with ADHD in a laboratory classroom setting.

DETAILED DESCRIPTION:
A single-center, dose-optimized, double-blind, randomized, placebo-controlled, parallel efficacy and safety laboratory classroom study with CTx-1301 in approximately 25 adults aged 18 to 55 years with ADHD. The study will be comprised of a screening period, a dose-optimization phase, a double-blind randomized phase, and a safety follow-up phase. Subjects will undergo a screening visit prior to entering a 5-week dose-optimization phase. During the dose-optimization phase subjects will have weekly visit and will be titrated to doses ranging between 25mg-50mg of CTx-1301. Eligible subjects will be randomized to their optimal dose or placebo in a 1:1 ratio after completing a practice Adult Laboratory Classroom (ALC) visit with 4 PERMP assessments. Subjects will take their assigned/randomized dose over the following 7-day period. On the 7th day subjects will complete a full ALC visit. The duration of the full ALC visit will be approximately 17 hours. Subjects will have an in-clinic safety follow-up visit within 7 days after the full adult laboratory classroom visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 55 years of age (inclusive) at the time of consent.
2. Subject must have a body mass index (BMI) ≥18.5 and ≤40.
3. Subject is unsatisfied with his/her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects who are naïve to pharmacological therapy for ADHD is permitted.
4. Negative serum beta-human chorionic gonadotropin (hCG) pregnancy test for subjects of child-bearing potential and must agree to remain abstinent or agree to use a highly effective, medically acceptable form of birth control for the time of written or verbal consent and for at least 30 days after the last dose of study drug has been taken (females) unless post-menopausal or surgically sterile. Male subjects with female partners must agree at Screening to remain abstinent or agree to use an effective and medically acceptable form of birth control from Screening to 90 days after the last dose of study drug.
5. Subject must be in general good health defined as absence of any clinically relevant abnormalities as determined by the Investigator based on physical and neurological examinations, vital signs, ECGs, medical history, and laboratory values (hematology, chemistry, or urinalysis) at Screening. If any of the exams or values are not within the laboratory reference range, the Investigator must review range and determine if clinically relevant. If clinically relevant, the subject is not eligible for the study.
6. Subject's intellectual function is at an appropriate level, as deemed by the Investigator.
7. Subjects need to be able to perform at least the basic level of problems on the PERMP pre-test with at least 10 questions answered correctly per page or 2 minutes performed at Visit 2.
8. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for the primary diagnosis of ADHD for any of the three presentations (combined, inattentive, or hyperactive/impulsive presentation) upon clinical evaluation and confirmed by the Mini International Neuropsychiatric Interview for Attention Deficit/Hyperactivity Disorder - Adults (MINI).
9. Subject must score 24 or higher on the Adult ADHD Investigator Rating Scale (AISRS) at the Screening visit (Visit 1) and Baseline visit (Visit 2) if no ADHD medication washout is required. For subjects requiring washout of ADHD medications, this criterion refers to a score following washout at the Baseline visit (Visit 2).
10. Subject must have a score of 4 (moderately ill) or higher on the clinician-administrated Clinical Global Impressions-Severity (CGI-S) scale at Screening. For subjects requiring washout of ADHD medications, this criterion refers to a score at the Baseline visit (Visit 2).
11. Subject must be able and willing to wash out of all stimulant ADHD medications (except study drug as indicated per protocol), including herbal medication, from 5 days prior to the start of the dose-optimization phase and for the duration of the entire study, defined as completion of the safety follow-up visit. Additionally, subject must be able and willing to wash out from all non-stimulant ADHD medications 21 days prior to the start of the dose optimization phase and for the duration of the entire study, defined as completion of the safety follow-up visit.
12. Subject must be able to read, write, speak, and understand English and be able to communicate with the Investigator and study coordinator in a satisfactory fashion and complete any study-related materials. Subject must plan to be available for the entire duration of the study.

Exclusion Criteria:

1. If female and of child-bearing potential, the subject must not be pregnant or breastfeeding at any time during the study or for 30 days following the completion of the study. If of child-bearing potential, urine hCG tests will be administered at protocol specified time points. Any positive pregnancy test during the study will exclude them from further participation in the study.
2. Subject has any psychiatric diagnosis of bipolar I or II disorder, current major depressive disorder, conduct disorder, disruptive mood dysregulation disorder, intellectual disability, obsessive-compulsive disorder, eating disorder, anxiety disorder (including generalized anxiety disorder), any history of psychosis, autism spectrum disorder, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances, or any other diagnosis/significant medical history that at the discretion of the Investigator excludes the subject from entry into the study.
3. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS-related disorders that might occur in childhood, or history of persistent neurological symptoms related to a serious head injury.
4. Subject has any clinically significant and/or unstable medical abnormality, chronic medical condition, persistent neurological symptoms, history of cardiovascular abnormality, abnormalities of respiratory, hepatic, gastrointestinal, renal, or any disorder or history of a condition that would impact or interfere with drug absorption, distribution, metabolism, or excretion during the study or may interfere with the participants ability to participate in the study.
5. Subject has family history of early cardiovascular disease or sudden death.
6. Subject has any history of attempted suicide or clinically significant suicidal ideation based on the Columbia Suicide Severity Rating Scale (C-SSRS) assessment, or answers "yes" to "Suicidal Ideation" item 4 or 5 in the past 3 years on the C-SSRS lifetime/recent assessment at Screening.
7. Subject has history of seizures, excluding febrile seizures.
8. Subject has a known primary sleep disorder (e.g., sleep apnea, narcolepsy, etc.)
9. Subject has a history of moderate to severe hypertension or has a resting sitting systolic blood pressure greater than140 millimeters of mercury (mmHg) or diastolic blood pressure greater than 90 mmHg.
10. Subject is considered treatment refractory by the Investigator.
11. Any use of anticonvulsants currently or within the past 2 years.
12. Uncontrolled thyroid disorder indicated by thyroid stimulating hormone (TSH) ≤0.8 x the lower limit of normal (LLN) or ≥ 1.25 x the upper limit of normal (ULN) from the reference laboratory.
13. Subject has first-degree relatives (biological parent or sibling) with a history of schizophrenia, schizoaffective disorder, bipolar I disorder, or bipolar II disorder.
14. Subject has history of substance abuse or shows evidence of substance or alcohol use disorder or has a positive urine alcohol or drug screen at Screening. Subjects with positive drug screens may be allowed to continue in the study if the result of the positive drug screen is from prescribed medications and the subject is willing to washout of the medication as required per protocol.
15. Subject has a history of physical, emotional, or sexual abuse resulting in a current diagnosis of posttraumatic stress disorder.
16. Previous treatment experience/exposure to CTx-1301.
17. Subject has a history of allergic reaction or sensitivity to methylphenidate, or any substance contained in CTx-1301 or the placebo drug.
18. Subject has participated in a laboratory study within 6 months prior to the start of Screening or has participated in any other clinical study with an investigational drug/product within 90 days prior to Screening or is currently participating in another clinical study.
19. Subject anticipates a move outside the geographic range of the investigative site during the duration of the study period or plans on travel that would not allow compliance to the protocol during the study period.
20. Subject is unsuitable in any other way to participate in the study, as determined by the Investigator.
21. Subjects who are family members of the employees at the study center, of the investigator, or those with direct involvement in the proposed study under the direction of that investigator or study center.
22. Subjects that live in the same household are not allowed to be in the same cohort.

Eligibility Criteria:

Subjects will be required to meet the following criteria at the end of the dose-optimization phase in order to be eligible for the double-blind, randomized treatment phase. These criteria are based on the efficacy and safety observed over the 5-week dose-optimization period.

1. A minimum of 2 sequential weeks on optimal dose.
2. A reduction of ≥ 30% of the AISRS from Visit 2 to Visit 7 during the dose optimization phase.
3. A CGI-I score of 1 or 2 points ("Very Much Improved" or "Much Improved") at the end of the dose optimization phase.
4. Acceptable tolerability of the optimized CTx-1301 dose during the dose optimization phase.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
The primary efficacy analysis will analyze the change in PERMP scores from Baseline (pre-dose) at Visit 8 to hour 16 at Visit 8. | Average of the change of the PERMP scores from baseline (measured pre-dose at Visit 8) to hour 16 at Visit 8.
  The Permanent Product Measure of Performance (PERMP) is an objective, validated, skill-adjusted math test that measures attention in ADHD. The PERMP total score comprises the sum number of math problems attempted and the number of math problems answered correctly. A higher PERMP score indicates lower impairment.

SECONDARY OUTCOMES:
Key secondary analysis will analyze the change in PERMP scores from baseline at each time point during the laboratory environment at Visit 8. | Baseline (pre-dose) at Visit 8 then post-dose at hours .5,1,3,6,9,12,13,14,15, and 16.
  The Permanent Product Measure of Performance (PERMP) is an objective, validated, skill-adjusted math test that measures attention in ADHD. The PERMP total score comprises the sum number of math problems attempted and the number of math problems answered correctly. A higher PERMP score indicates lower impairment.
Key secondary analysis will analyze the change from baseline (pre-dose at Visit 2) of Clinical Global Impression - Severity (CGI-S) scores to CGI-S at Visit 8. | Baseline (pre-dose at Visit 2) to Visit 8 (approximately 6 weeks).
  The CGI-S is a single score ranging from 1-7; an improvement from Baseline is defined as a decrease in the score.

OTHER OUTCOMES:
Safety - incidence of TEAEs | Screening (Visit 1) to Visit 9 (approximately 7-11 weeks, depending on screening window)
  Treatment Emergent Adverse Events (TEAEs) will be evaluated at each visit
Safety - incidence of changes in vital signs, BMI, blood labs, physical exams, Columbia-Suicide Severity Rating Scale (CSSR-S), and ECGs. | Screening (Visit 1) to Visit 9 (approximately 7-11 weeks, depending on screening window)
  Safety will be assessed at each visit. Any clinically significant changes will be reported as an adverse event.
Exploratory endpoints will evaluate the efficacy of CTx-1301 during the dose optimization phase. | Screening (Visit 1) to Visit 7 (approximately 6-10 weeks, depending on screening window).
  Evaluate overall treatment experience of subjects who were stable on ADHD stimulant medications within the 30 days prior to Screening at Visit 1 compared to CTx-1301 at the end of the dose optimization phase by utilizing the provided prior medication entrance questionnaire and the existing medication exit questionnaire.
The purpose of this study is to estimate the effect size of treatment on the PERMP instrument in an adult ADHD population as defined by the inclusion/exclusion criteria. | Screening (Visit 1) to Visit 9 (approximately 7-11 weeks, depending on screening window)
  The purpose of this study is to estimate the effect size of treatment on the PERMP instrument in an adult ADHD population as defined by the inclusion/exclusion criteria.Though primary and secondary endpoints are defined in accordance with International Conference on Harmonization (ICH) E9 guidelines, this study is not intended to demonstrate statistical significance via treatment group comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Principal Investigator
Locations (1):
- Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada, United States